CLINICAL TRIAL: NCT06213272
Title: Improving Reading Competence in Aphasia With Combined Aerobic Exercise and Phono-Motor Treatment
Brief Title: Combined Exercise and Targeted Therapy for Post-Stroke Reading Deficits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Olga Boukrina, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-1242-23
Record Dates: First submitted 2023-12-26; First posted 2024-01-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Aphasia; Reading Disorder
Keywords: exercise; stroke; aphasia; reading therapy; phono-motor therapy; aerobic exercise treatment; MRI
MeSH Terms: conditions — Stroke; Aphasia; Dyslexia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the 2 intervention groups: combined aerobic exercise and phono-motor therapy, or combined light stretching and phono-motor therapy. Randomization will be stratified by aphasia severity.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will not be informed about study hypotheses. Outcome Assessors will be masked to participants' assigned condition. Treating therapists (care providers) will be masked to participants baseline and outcome scores.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Exercise Treatment (AET) combined with Phono-Motor Therapy (PMT) (Experimental): Patients will receive 40, once-daily 2-hour intervention sessions administered 4-5 times per week by trained research assistants. Sessions will begin with a 5-min warm-up, followed by 20 min of aerobic exercise (cycling, 60% heart rate range), and a 5-min cool-down. Participants will rate their perceived effort every 5 minutes and complete a log at the end of each session to characterize their experience. When HR returns to near resting levels (i.e., 5-min after cool-down), participants will undertake the PMT for the remaining 90 min.
  Interventions: Behavioral: Phono-Motor Therapy; Behavioral: Aerobic Exercise Training (AET)
- Stretching and PMT (Active Comparator): Patients will receive 40, once-daily 2-hour intervention sessions administered 4-5 times per week by trained research assistants. Sessions will begin with a 5-min warm-up, followed by 20 min of stretching and a 5-min cool-down. Stretching activities will target the head/neck, shoulder, elbow/forearm, hand/wrist, trunk/hip, ankle/foot. Participants will complete a log at the end of each session to characterize their experience, and within 5 min of completing the last stretching activity, participants will undertake PMT for the remaining 90 min of a given session.
  Interventions: Behavioral: Phono-Motor Therapy; Behavioral: Stretching

INTERVENTIONS:
Behavioral: Phono-Motor Therapy — The goal of PMT is to build orthographic and phonological awareness and phonological sequence knowledge. During PMT, participants will complete a series of tasks manipulating minimal sound units (consonants (C) & vowels (V)), combining these units into syllables (CVC, CVCC, CCVC) and syllable sequences (real words and readable nonwords). PMT will aim to engage 5 modalities: visual, acoustic, tactile kinesthetic, motor, and orthographic. Multisyllabic stimuli used during treatment will consist of 40 real words and 68 readable nonword letter strings.
Behavioral: Aerobic Exercise Training (AET) — Stationary ergometer cycling at 60% heart rate range for 20 minutes, plus 5 minutes of warm up and cool down.
  Arms: Aerobic Exercise Treatment (AET) combined with Phono-Motor Therapy (PMT)
Behavioral: Stretching — Light stretching activities targeting the head/neck, shoulder, elbow/forearm, hand/wrist, trunk/hip, ankle/foot.
  Arms: Stretching and PMT

SUMMARY:
The goal of the proposed project is to test the effectiveness of a novel hybrid approach to treatment of reading disorders after stroke, in which exercise training will be used in combination with a targeted reading treatment. This approach is expected to increase cerebral circulation and help to rebuild and strengthen the damaged phonological neural networks. Through this combinatory approach, the study aims to enhance the reading and language improvements seen with existing treatments.

DETAILED DESCRIPTION:
Close to 2.5 million Americans are currently living with post-stroke aphasia, a debilitating communication disorder affecting multiple language modalities. Most stroke survivors with aphasia have acquired reading deficits, which persist chronically and severely limit life participation and autonomy. There is an urgent need for effective treatments grounded in stroke neurobiology which yield robust functional improvements. This project is a randomized controlled trial, which will recruit 70 individuals with chronic left-hemisphere stroke. Participants will complete 40 sessions of targeted reading treatment combined with either 20 minutes of moderate aerobic exercise or light stretching. Participants will undergo 3 Magnetic Resonance Imaging (MRI) scans, administered before the intervention, after the initial exercise session, and after the full course of treatment. They will also complete behavioral testing before and after the intervention. The outcome of this study has the potential to radically change how reading treatments are applied, increasing their effectiveness, and ultimately improving the lives of 2.5 million Americans living with stroke-related aphasia. In addition, it is likely that the results will contribute to the understanding of stroke recovery mechanisms thereby fundamentally advancing the field of neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* fluent and literate in English prior to stroke
* 1st ever stroke
* more than 3 months post-stroke
* post-stroke reading deficits, defined as reading aloud accuracy <83% for single words or <65% for readable nonwords
* living within a 50-mile radius from Kessler Foundation.

Exclusion Criteria:

* contraindication to MRI
* prior neurological disease
* developmental learning or reading disability (i.e., developmental dyslexia)
* contraindication to exercise
* concurrent speech and language therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Reading Aloud | Baseline and within 2 weeks of treatment completion (~10 weeks from study onset)
  Participants will read aloud 120 words and 80 nonwords, some of which will be selected for PMT based on individual accuracy (treated items). A subset of these will not be treated and will be used to assess generalization.
2 Alternative Forced Choice Computer Tasks | Baseline and within 2 weeks of treatment completion (~10 weeks from study onset)
  Touch-screen computer tests of semantics, phonology, & orthography (composite score).
  Participants choose one of two examples on the screen that matches a target in meaning (semantics), rhymes with the target (phonology), or chose a letter string that more closely resembles a word.
Reading Comprehension Battery for Aphasia - 2nd edition (RCBA-2) | Baseline and within 2 weeks of treatment completion (~10 weeks from study onset)
  Letter, word, sentence, paragraph, and text-level reading comprehension test for aphasia.
Cerebral Blood Flow (CBF) | Baseline, after a single session of acute exercise, and within 2 weeks of treatment completion (~10 weeks from study onset)
  CBF will be measured using an Arterial Spin Labeling MRI sequence
Resting State Functional Connectivity (rsFC) | Baseline, after a single session of acute exercise, and within 2 weeks of treatment completion (~10 weeks from study onset)
  RsFC will be measured using fMRI acquired with rapid simultaneous multi-slice echo-planar imaging (EPI) (TR=1.5s, TE=30ms, 44 slices, gap = .5mm, 2mm isotropic voxels, N volumes=400, eyes open). To standardize the rest condition across participants, we will instruct participants to look at a centrally presented fixation dot for the duration of the scan.
Task-induced fMRI activation | Baseline and within 2 weeks of treatment completion (~10 weeks from study onset)
  Data will be collected using fMRI sequence above. Participants will perform a reading aloud task where words or nonwords are presented on the screen one at a time. The order of reading blocks (words/nonwords) will be randomized (9 blocks of each*2 runs). Each 32 s reading block will have 8 words (blocked by condition, e.g., high imagery, frequency, and consistency) or nonwords, presented for 1 s and followed by ~3s response period. The onset of each word or nonword stimulus will be randomly jittered by 100-400ms to provide the ability to model errors. Voice responses will be collected via an MR microphone (FOMRI III+, Optoacoustics) and used to score reading accuracy. Reading aloud accuracy will be evaluated by 2 independent raters, and disagreements will be resolved by discussion. The reading aloud blocks will be alternated with baseline fixation blocks (12s) and rest blocks (8s) for a total duration of 52s for each block cycle (7.8 min run)

SECONDARY OUTCOMES:
Western Aphasia Battery Revised | Baseline and within 2 weeks of treatment completion (~10 weeks from study onset)
  A comprehensive assessment of language impairments in aphasia
Philadelphia Naming Test (Short) | Baseline and within 2 weeks of treatment completion (~10 weeks from study onset)
  A 30-tem picture naming test designed to identify word finding difficulties. It is presented on a computer using line drawn images of animate and inanimate objects and is audio recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Boukrina, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
The scientific data and metadata generated by this project will be securely archived in several repositories. Our study design will be hosted on ClinicalTrials.gov, the code will be stored on GitHub, and the neuroimaging data alongside behavioral datasets will be deposited on OpenNeuro.org. Each repository will contain links to the others, ensuring seamless accessibility and discoverability of all associated data and metadata across the platforms.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Data sharing will occur no later than the time of an associated publication of primary study outcomes or 1 year from the end of the performance period, whichever comes first.
  Data stored in repositories such as OpenNeuro.org, GitHub, and ClinicalTrials.gov are typically retained long term, often without a predetermined deletion date. Therefore, barring any unforeseen changes to these platforms' policies, the data from this project will be available for an indefinite period of time, allowing scientific community to access and utilize the available information.
Access Criteria: Access to the scientific data will require users to create an account with the respective repository (GitHub or OpenNeuro.org). After this step, they will be able to freely access and use the data, following the repository's terms of use. Study design data, which will be hosted on ClinicalTrials.gov, will be available to users without registration.
URL: http://OpenNeuro.org